CLINICAL TRIAL: NCT00870701
Title: Randomised Multicentric Phase III Study Comparing Observation Versus Post-surgery Radiotherapy After Complete Exeresis With Margins Greater Than or Equal to 1 cm in Soft Tissues Members Sarcoma.
Brief Title: Observation Versus Post-surgery Radiotherapy After Complete Exeresis in Soft Tissues Members Sarcoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08SARC01
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Soft Tissue Sarcoma of Members
Keywords: sarcoma; soft tissue; members; radiotherapy; absence of radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absence of Radiotherapy (Experimental): No Radiotherapy; Simple monitoring without active treatment
  Interventions: Other: absence of radiotherapy
- Radiotherapy (Active Comparator): Radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — 50 grays in 25 fractions of 2 Gys or 50.4 grays in 28 fractions of 1.8 grays
  Arms: Radiotherapy
Other: absence of radiotherapy — absence of radiotherapy
  Other Names: Simple monitoring; Observation
  Arms: Absence of Radiotherapy

SUMMARY:
Soft tissue sarcomas represent less than 1% of malignant tumors in adults and sarcomas members represent 60% of them.

These rare tumors involve complex multidisciplinary care better in centers having expertise.

Loco-regional therapy strategies have evaluated over time for tumors of members leading to propose more often the combination of a large conservative tumor excision with radiotherapy. Results have been demonstrated equivalent to those of an amputation in terms of local control and survival.

The local recurrence rate for sarcomas of the members of any kind after surgery with or without radiotherapy in the literature varies from 10 to 30%.

The main objective is to achieve a low recurrence rate while maintaining the function. The question remains the possibility of an absence of irradiation in selected cases in a de-escalation therapy order.

ELIGIBILITY:
Inclusion Criteria:

* Soft tissue sarcoma members histologically confirmed
* Tumor primitive complete excision with margins greater than or equal to 10 mm in the soft tissue in all directions during the initial surgery.

A sub-centimeter margin is authorized under an anatomic barrier (fascia, fascia, inter-osseous membrane, periosteum), if surgery is R0 a margin sub-centimeter depth is allowed for superficial tumors if the underlying fascia RESECTED is not invaded.

* Primitive tumors without breaking initial tumor and without tumor residue in the systematic recovery in case of incomplete initial excision margins or doubtful
* WHO less than or equal to 2
* Age greater than or equal to 18 years
* Review extension negative (normal chest CT)
* Information and monitoring possible
* Patient affiliated to social security

Exclusion Criteria:

* Previously treated local sarcoma relapse
* Visceral or lymph node metastases
* pre-operative treatment (chemotherapy or radiotherapy)
* PNET, alveolar rhabdomyosarcoma, Darrier-Ferrand sarcoma
* excision margins of less than 10 mm in one direction or doubtful or unspecified, except under an anatomic barrier (fascia, fascia, inter-osseous membrane, periosteum), if surgery is R0 and tumors if the superficial fascia underlying RESECTED is not invaded.
* Break-tumor during the initial surgery, or residual tumor at second surgery
* Chemotherapy
* Delay between surgery R0 margins greater than or equal to 1 cm (initial surgery or recovery) and the start of radiotherapy exceeding 8 weeks
* History of radiation on the Member
* History of cancer (except carcinoma in situ of the cervix and basal cell skin cancer or in complete remission for over 5 years)
* Pregnant Women
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-03-19 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of local control at 5 years after surgery compared with exclusive post-operative radiotherapy for soft tissue tumors of the members who have surgery with wide excision margins greater than or equal to 10 mm. | 2021

SECONDARY OUTCOMES:
Evaluation of the quality of life by questionnaire of quality of life QLCQ30 | 2021
Evaluation of acute and late complications | 2009 to 2021
Overall Survival | 2021

CONTACTS AND LOCATIONS:
Overall Officials: Martine DELANNES, MD, Principal Investigator — Institut Claudius Regaud
Locations (18):
- France (18):
  - Institut de Cancérologie de l'Ouest - Centre Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Mondor, Créteil
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU de la Timone, Marseille
  - Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier
  - Centre Alexis Vautrin, Nancy
  - Centre Antoine Lacassagne, Nice
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest - Centre René Gauducheau, Saint Herblain (Nantes)
  - Institut de Cancerologie de La Loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif